CLINICAL TRIAL: NCT04406233
Title: Muscle Mass and Strength as Predictors of Time to Medical Discharge and Mortality in Patients Hospitalized With COVID-19: A Prospective Observational Study
Brief Title: Muscle Mass and Strength as Predictors of Time to Discharge in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Phd, University of Sao Paulo
Other Study IDs: 31303720.7.0000.0068
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The severe acute respiratory syndrome induced by the new coronavirus (SARS-CoV-2) has been declared a worldwide pandemic. Identifying common characteristics of the disease is crucial to promote a better prognosis for patients and to reduce the occurrence of medical complications, the time to medical discharge and mortality rates. Muscle mass and strength are recognized predictive measures of medical complications and mortality in different populations, but it is still unclear whether these also applies to patients with SARS-CoV-2. Therefore, this study will investigate whether muscle mass and/or muscle strength are predictors of the time until medical discharge of patients hospitalized with SARS-CoV-2. Our working hypothesis is that muscle mass and/or muscle strength are predictive measurements of the time until medical discharge of patients hospitalized with SARS-CoV-2

DETAILED DESCRIPTION:
Muscle mass (via ultrasound) and muscle strength (via handgrip) of patients with SARS-CoV-2 will be assessed upon admission, medical discharge and 180 days after medical discharge. The time until medical discharge and any medical complications will be recorded. Throughout the hospitalization period, the mortality rate will also be assessed. One hundred and eighty days after medical discharge, the number of hospital readmissions, mortality rate and the use of public health services will be evaluated, to estimate the cost of each patient to the health service. Patients will be stratified according to muscle mass and strength assessed at admission. Data will be analysed using a mixed model with repeated measures assuming group (percentiles) and time (admission, medical discharge, and 180 days after medical discharge) for each dependent variable. In the event of a significant F-value, Tukey-Kramer post hoc adjustments will be used for multiple purposes. Survival rate will be examined using the Kaplan-Meier curve and analyzed using the Log-rank test (Mantel-Cox). The level of significance will be set apriori at P≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older ;
* hospital stay less than 48 hours;
* length of hospital stay to 48 hours no requiring invasive mechanical ventilation;

Exclusion Criteria:

* cancer in the last 5 years;
* delirium;
* cognitive deficit that impossibility the patient to read and sign the informed consent form;
* neurological disease;
* degenerative muscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2020-05-23 (Actual); Primary Completion 2022-05-23 (Estimated); Study Completion 2022-05-23 (Estimated)

PRIMARY OUTCOMES:
Time to medical discharge | through the hospitalization period, an average of 15 days
  Length (in days) of the time hospitalization until medical discharge

SECONDARY OUTCOMES:
All-cause mortality | through the hospitalization period, an average of 15 days, 60, 180 and 360 days after medical discharge
  All-cause mortality rate along the study
Hospital readmission | 60, 180 and 360 days after medical discharge
  Occurrence of medical complications that require hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Univsersity of Sao Paulo, São Paulo, Brazil